CLINICAL TRIAL: NCT02820090
Title: The Predictive Effect of the Inflammatory Response on the Evacuation of Mechanical Ventilation and the Mechanism
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Yingmin Ma, Vice President of the Beijing Chao Yang Hospital, Beijing Chao Yang Hospital
Other Study IDs: 15210511726
Record Dates: First submitted 2016-05-31; First posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Systemic Inflammatory Response Syndrome; Ventilator Weaning
Keywords: Inflammatory Factor; Mechanical Ventilation
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Success with SBT: The patient have a success in SBT.
- Success with mechanical ventilation: Weaning from mechanical ventilation is successful
- failure with SBT: The patient have a failure in SBT.
- failure with mechanical ventilation: Weaning from mechanical ventilation is failed

SUMMARY:
Infection and trauma take a important role in the acute respiratory failure.There are different causes and degrees of inflammatory reaction in the critically ill patient. The inflammatory reaction should also affect patients on mechanical ventilation dependence with body physiological response and disease prognosis in patients. Therefore, the investigators hypothesize that inflammation may have an important role in the prediction of weaning from mechanical ventilation.

DETAILED DESCRIPTION:
In the process of mechanical ventilation, the patients were divided into two groups according to the failure of spontaneous breathing test and spontaneous breathing test.In the index of predicting mechanical ventilation, the investigators will take the index of inflammatory response, the function index of diaphragm and the amount of exhaled CO2 into account to reduce the failure rate of mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* oral, nasal tracheal intubation and mechanical ventilation in patients with respiratory failure
* mechanical ventilation time over than 48 hours
* Glasgow score greater more than or equal to 13 points

Exclusion Criteria:

* Aged less than 14 years or more than 80 years old
* patients with neuromuscular disease
* pure heart failure pulmonary edema patients
* patients with tracheotomy

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patient with oral or nasal tracheal intubation and mechanical ventilation in respiratory failure
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
The relationship between mechanical ventilation of ventilator and inflammatory response | January 2014 to December 2016
  Through the study of mechanical ventilation weaning success and failure of patients with respiratory physiological indicators, blood, urine related inflammatory indicators, analysis of the relationship between inflammatory response and mechanical ventilation weaning.The test indicators include C- reactive protein, tumor necrosis factor and some interleukin for related.

SECONDARY OUTCOMES:
The relationship between diaphragm movement function and weaning from mechanical ventilation | January 2016 to December 2017
  To study the relationship between the inflammatory response and the contractile function of diaphragm, which is helpful to judge the effect of inflammatory factors on the evacuation of mechanical ventilation.
the output of CO2 | January 2016 to December 2017

CONTACTS AND LOCATIONS:
Overall Officials: MA yingmin, professor, Study Director — Beijing Chao Yang Hospital

IPD SHARING:
Plan to Share IPD: Yes